CLINICAL TRIAL: NCT04427436
Title: Investigating the Potential of Novel Dementia Biomarkers - an MRI, fNIRS and EEG Study
Brief Title: Novel Dementia Biomarkers
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: German Center for Neurodegenerative Diseases (DZNE) (Other)
Collaborators: Otto-von-Guericke University Magdeburg (Other)
Responsible Party: Principal Investigator, Notger Müller, Professor Dr. Notger Müller, German Center for Neurodegenerative Diseases (DZNE)
Other Study IDs: MD070
Record Dates: First submitted 2020-05-14; First posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Alzheimer Disease, Early Onset
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Mild Cognitive Impairment (clinical determination)
  Interventions: Other: No Intervention
- Control: Healthy Elderly
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No Intervention

SUMMARY:
The study will investigate structural and functional characteristics of the brain of dementia patients compared to healthy controls in order to get a better insight into importance of early biomarkers for the diagnosis of Alzheimer's dementia. The methods for obtaining biomarkers incude magnetic resonance imaging (MRI), near-infrared spectroscopy (fNIRS) and electroencephalography (EEG), electrocardiography (ECG) and neurophyshological assessments. Special parameters are being studied that have already been shown to detect changes in the early stages of Alzheimer's dementia.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed MCI patients and matched healthy controls

Exclusion Criteria:

* Metal in body and tatoos;
* Other chronic systemic neurological, cardiologic, metabolic or musculo-skeletal diseases which have been proven to influence the outcome variables
* Alcohol abuse
* Colour blindness
* Pregnancy
* Surgery in the last 6 months
* Uncorrected vision

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients aged between 50 and 80 years will be recruited from the memory clinic at the Department of Neurology of the Otto von Guericke University Clinic, Magdeburg, Germany. The diagnosis of MCI/AD will be established by experienced neurologists of the memory clinic according to standardised criteria. Control participants will be matched by education, age and gender. These will be recruited through advertisement.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Locus Coeruleus (LC) Intensity | 15 minutes
  LC-intensity can be assesed with specific MRI sequences (TSE MRI-Sequence (see Dordevic et al, 2017))
Volume of brain regions | 30 minutes
  VBM (voxel-based morphometry)
fNIRS-based change in oxyhemoglobin and deoxyhemoglobin | 1 hour
  In response to each task there is a hemodynamic response, which can be measured by fNIRS. In particular, fNIRS measures changes in blood oxy- and deoxy-hemoglobin.
Event-related-potential (ERP) waveforms: negative deflections (N100, N300) and positive deflections (P100, P300) | 1 hour
  Voltages generated in the brain structures in response to specific events (Event-related potentials (ERPs))
Heart Rate Variability (HRV) | 1 hour
  ECG-based variability measures in R-R intervals, both in rest abd during tasks
Score on CERAD-Plus | 30 minutes
  Cognitive performance measure in points, with a higher score meaning better performance
Error-rate on Stroop-test | 10 minutes
  Test of executive functions, higher error-rate means worse performance
Error-rate on N-Back-test | 10 minutes
  Working memory test, higher error-rate means worse performance
Performance on verbal fluency test | 10 minutes
  Test of verbal fluency, more words spoken means a better score

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Grassler B, Herold F, Dordevic M, Gujar TA, Darius S, Bockelmann I, Muller NG, Hokelmann A. Multimodal measurement approach to identify individuals with mild cognitive impairment: study protocol for a cross-sectional trial. BMJ Open. 2021 May 25;11(5):e046879. doi: 10.1136/bmjopen-2020-046879. PMID 34035103